CLINICAL TRIAL: NCT03412058
Title: Prospective Cohort Study to Identify the Predictive Factors of Response to PD-1 or PD-L1 Antagonists
Brief Title: Identifying the Predictive Factors of Response to PD-1 or PD-L1 Antagonists
Acronym: CHECK'UP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UC-0108/1708
Record Dates: First submitted 2017-11-14; First posted 2018-01-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: PD-1; PD-L1
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Melanoma (Experimental): Biopsy and blood samples will be collected from patients treated with an antiPD-1 or antiPD-L1 antibody with marketing authorization for the indication, during the course of their treatment
  Interventions: Procedure: Biopsy
- NSCLC (Experimental): Biopsy and blood samples will be collected from patients treated with an antiPD-1 or antiPD-L1 antibody with marketing authorization for the indication, during the course of their treatment
  Interventions: Procedure: Biopsy
- HNSCC (Experimental): Biopsy and blood samples will be collected from patients treated with an antiPD-1 or antiPD-L1 antibody with marketing authorization for the indication, during the course of their treatment
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — To be performed prior to anti-PD1/PD-L1 treatment initiation
Procedure: Biopsy — To be performed after 42 (±3) days of anti-PD1 or PD-L1 treatment in consenting patients
Procedure: Biopsy — To be performed at disease progression if medically feasible

SUMMARY:
This is a prospective cohort study which aims to identify predictive factors of response to PD-1 and PD L1 antagonists authorised for use in France in treatment of melanoma, NSCLC, or HNSCC.

DETAILED DESCRIPTION:
The study will include 670 patients with melanoma, NSCLC, or HNSCC who are set to receive treatment with a single-agent PD-1 or PD L1 antagonist regimen as indicated in the respective European MA or under the conditions of a TAU and according to the standard practices at the investigational site.

Included patients will be followed for a total of 5 years. Prior to initiation of PD-1 or PD-L1 antagonist therapy, included patients will undergo a biopsy of a tumour lesion (unless suitable archived material is available) and provide a blood sample for immunohistochemistry and genomic studies. Patients at selected participating sites will also be asked to provide stool and saliva samples (optional). Additional optional biopsy samples may be collected from consenting patients after 42 (±3) days of PD-1 or PD-L1 antagonist treatment and in the event of disease progression or recurrence. Additional blood samples will also be collected at regular intervals throughout the observation period until disease progression, regardless of whether PD-1 or PD-L1 antagonist treatment is ongoing or has discontinued. Efficacy of treatment will be evaluated using both Response Evaluation Criteria in Solid Tumours (RECIST) and immune-related RECIST (iRECIST). Information regarding the PD-1 or PD-L1 antagonist related toxicities, subsequent antineoplastic treatments, and survival status will also be collected during the trial.

An elastic-net approach will be used to identify correlations between different parameters and develop a signature of response to treatment. For each indication, the patients will be separated into two cohorts: a 'training' cohort and a 'validation' cohort. The 'training' cohort will be made up of the first patients included in the indication and will be used to develop a predictive response score. The 'validation' cohort will include all the remaining patients. The performance of the predictive score will be tested in this second cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Histological confirmed diagnosis of one of the following:

   * Non-resectable (stage III) or metastatic (stage IV) melanoma,
   * Metastatic, EGFR- and ALK-negative, non-small cell lung cancer with a high level of PD-L1 expression (defined as a "tumour proportion score" of greater than or equal to 50%) which has not been previously treated with chemotherapy in the metastatic setting,
   * Head and Neck squamous cell carcinoma that is that is recurrent or progressing following reference chemotherapy and that is not amenable to surgery or radiation therapy.
3. Indicated for treatment with a PD-1 or PD-L1 antagonist according to the European Marketing Authorisation or the conditions of a Temporary Authorisation of Use.
4. Estimated life expectancy ≥16 weeks.
5. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.
6. Presence of at least one tumour lesion (except bone lesions) accessible to biopsy, if a biopsy is required (see below).
7. Willing and able to provide a pre-treatment biopsy sample, if a biopsy is required.

   Note: where an archived tumour sample is available, this archived sample can be used in place of a fresh biopsy sample, if the patient has not received any antineoplastic therapy since the collection date.
8. Measurable disease according to RECIST v1.1 (Eisenhauer, 2009).
9. Beneficiary of social insurance coverage.
10. Comprehension of French.
11. Provision of written informed consent (signed and dated) prior to the initiation of any protocol specific procedure.

Exclusion Criteria:

1. Any contraindication to treatment with a PD-1 or PD-L1 antagonist.
2. Any contraindication to a biopsy including: platelets <80 x 10⁹/L, International Normalised Ratio (INR) >1.5 or prothrombin time (PT) >1.5 x upper limit of normal range (ULN), prolonged partial thromboplastin time (PTT) in the absence of factor XII deficiency or antiphospholipid antibodies, ongoing treatment with anticoagulants.
3. Bone metastasis as the only disease site available for biopsy.
4. Previous treatment with a PD-1 or PD-L1 antagonist.
5. Individuals deprived of liberty or placed under the authority of a tutor.
6. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of response signature | 84 days
  The sensitivity is defined as the ratio of patients classified as responder by the signature to the number of patients presenting an objective response (CR or PR) according to centralized assessment of RECIST v1.1.

SECONDARY OUTCOMES:
Frequency and severity of adverse events occuring during the observation period | Through treatment period
  Adverse events will be evaluated according to NCI-CTCAE v4
Objective response | 84 days
  Objective response as assessed by Investigators according to RECIST v1.1.
Objective response | 84 days
  Objective response as assessed centrally according to RECIST v1.1.
Progression-free survival | 5 years
  defined as the time from inclusion until documented disease progression (PD) according to RECIST v1.1, or death, whichever occurs first.
iProgression-free survival | 5 years
  defined as the time from inclusion until documented PD according to iRECIST or death, whichever occurs first.
Overall survival | 5 years
  defined as the time from inclusion until death due to any cause.
Duration of response | 5 years
  defined as the time from first observation of objective response according to RECIST v.1.1 until PD or death, whichever occurs first
Treatment costs | 5 years
  including cost of antiPD-1/PD-L1 treatment and supportive care for antiPD-1/PD-L1 treatment-related adverse events
Tumour size | 5 years
  Changes in tumour size over time

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Penault-Llorca, Principal Investigator — Centre Jean Perrin
Locations (19):
- France (19):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Caen, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Inter. de Creteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut de cancérologie de l'ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - CHU Saint-Etienne, Hôpital Nord, Saint-Etienne
  - Institut Claudius Regaud - IUCT- 0, Toulouse
  - CHU de Tours, Tours
  - Institut Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif